CLINICAL TRIAL: NCT05047432
Title: Concordance Of Methods to Select Tracheostomy Tube Size for Adults in Intensive Care
Acronym: COMETS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 136601; 272157 (Other: Integrated Research Application System (UK)); NIHR300537 (Other Grant/Funding Number: National Institute for Health Research (UK))
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Tracheostomy
Keywords: tracheostomy; tracheotomy; trachea; biometrics
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional trial — Non-interventional trial

SUMMARY:
This study is part of a larger PhD project. The aim of the overall project is to provide evidence to help healthcare staff choose the best size tracheostomy breathing tube for patients in intensive care. There are no clear guidelines on how to choose the size of tracheostomy tubes currently.

The aim of this part of the project is to compare methods of choosing the size tracheostomy tube for patients. Four methods are based on easily recorded physical characteristics of the participants (sex, height, Body Mass Index and shoulder width). A fifth method is based on measurement of the windpipe (trachea). We will recruit patients and staff at the Royal Free London NHS Foundation Trust. We will measure their height, weight and shoulder width, and record their age and sex. We will use ultrasound to measure each participant's trachea.

We will calculate the recommended tube size using the five methods above. We will compare how well the first four methods agree with the method based on measurements of the trachea.

The results of this study will inform healthcare staff how well the different ways of choosing the size of tube relate to the fit of a tube in the trachea.

DETAILED DESCRIPTION:
1. INTRODUCTION This piece of research constitutes one of four workstreams in an NIHR funded PhD programme of work. The overall aims of the PhD project are 1) to create guidance for Health Care Professionals (HCPs) on how to select the right size tracheostomy tube (TT) for patients in an intensive care unit (ICU), and 2) to identify ways to best ensure that HCPs follow the guidance.

   This protocol is for Workstream 2. In this workstream we will calculate tube size recommendations for each participant using five methods:
   * four using sets of criteria that replicate current practice and relate to physical characteristics (sex, shoulder width, height and Body Mass Index)
   * a recommended set of criteria based on measurements of tracheal width

   We will then calculate concordance (%) between tube size recommendations based on tracheal measurements and those based on other physical characteristics. Secondary analysis will determine strength of correlation between tracheal diameter and height, shoulder width, age, sex, Body Mass Index and ethnicity. The findings will provide evidence for clinicians on how the fit of a tracheostomy tube within the trachea may be affected by the size-selection criteria used.

   This study in isolation is not intended to provide definitive clinical recommendations regarding the selection of tracheostomy tube size, since this also requires knowledge of 1) the impact of tube size on airflow through and around tracheostomy tubes and 2) what is important to patients in terms of functional effects of size of tube. These two issues are the focus of other workstreams within the larger programme of work.
2. BACKGROUND AND RATIONALE

   Tracheostomy tubes (TT) are breathing tubes that are surgically inserted through the front of the neck. They can:
   * allow easier breathing for patients with upper airway obstruction
   * provide access to the lungs to clear secretions
   * facilitate longer term use of artificial breathing machines (mechanical ventilation, MV) by replacing breathing tubes that go through the mouth
   * help patients to be liberated from MV There are an estimated 12,000 tracheostomy insertions a year in England and the majority of these occur in intensive care units (ICUs). There are a number of widely used reference guidelines addressing the general management of patients with a TT. These state that a clinician should consider the size of the TT prior to insertion, but do not fully describe how to select the correct size. In practice, methods of selecting tracheostomy tube vary widely and decisions are often made on the basis of a patient's sex or perceived size.

   TTs that are the wrong size can cause physical and psychological harm. If the TT is too small there is a risk of a leak around the tracheostomy cuff (a ring-shaped balloon around the tube), leading to difficulty using MV, and aspiration of saliva or stomach contents into the lungs. Over-inflation of TT cuff in an attempt to compensate for the TT being too small can cause long-term damage to the trachea. If the TT is too big there is risk of trauma to the skin around the hole in the neck and to the trachea, and a patient is unlikely to be able to use a speaking valve to talk. In TTs that are too big or small, the tip may abut the anterior or posterior tracheal wall, causing trauma and difficulty breathing around or through it respectively. Any trauma to the tracheal wall or insertion site can lead to narrowing of the airway called tracheal stenosis. The consequences of this range from mild breathing difficulties through to complete blockage of the airway. Treatment for tracheal stenosis ranges from balloon dilatation to major reconstructive surgery and can cause a heavy burden to patients and the health services. Good decision-making regarding size of TT may reduce the incidence of tracheal stenosis and associated financial costs of treatment or increased levels of care.

   If the TT is too big, a patient is unlikely to be able to talk. Not being able to talk is highly stressful for patients on ICU. It can lead to treatment decisions being delayed or made by others on behalf of the patient, and has been linked with increased levels of anxiety and depression and the development of delirium and post-traumatic stress disorder.

   There is mixed evidence to support correlation between anthropometrics and tracheal dimensions. A few observational cohort studies have sought to establish normative data for tracheal dimensions, some comparing these with sex, height, or weight. Evidence from a paediatric study supports a correlation between height and tracheal dimensions in children. The literature on adults is inconclusive. No studies to date have investigated a potential correlation between shoulder width and tracheal diameter. Tracheal width in men, like shoulder width, continues to grow beyond the point when full stature is achieved, and has been proposed as a cause for a non-linear relationship between height and tracheal width found in some studies. 'Patient size' is commonly used in tracheostomy tube decisions. Height, shoulder width and BMI are used in this study as surrogates for patient size.

   Ultrasound is increasingly being used to assess the airway and has shown strong correlation with measurements taken from computed tomography (CT) and magnetic resonance imaging (MRI). Ultrasound has the benefits over other measurement techniques of being non-invasive, not requiring radiation exposure and being relatively inexpensive.
3. OBJECTIVES 3.1 Primary Objective To determine the concordance between a tracheal diameter-based standard for selecting tracheostomy tube size and sets of criteria based on sex, height, shoulder-width and BMI in an adult population.

   3.2 Secondary Objectives To estimate the association between tracheal width and standing height, shoulder width, ethnicity, age, sex and other demographic characteristics in an adult population.
4. STUDY DESIGN Type of Study: cross-sectional observational study Population: Adult inpatients, outpatients and hospital staff at the Royal Free London NHS Foundation Trust. Prisoners, patients and staff who are pregnant, those with severe deformity of the spine and patients lacking mental capacity to consent will be excluded.

   Duration of enrolment: One appointment of 45-60 minutes. No follow-up required. Sample size: a sample of 114 participants will provide 90% power to detect a concordance of 65% (null hypothesis = 50%) between methods of selecting tracheostomy tube size, with a 1-sided significance level of 2.5%.

   Statistical Analysis: Analysis of concordance will be used to evaluate the level of agreement between methods to select size of tracheal tube using 1. tracheal width as measured using ultrasound 2. other physical characteristics (sex, height, shoulder width, BMI) Concordance will be expressed as proportion (%) of agreement. Univariate and multivariate linear regression analysis will be used to evaluate the association between tracheal width and standing height, shoulder width, ethnicity, age, sex and other demographic characteristics.
5. STUDY SCHEDULE We will advertise the study via flyers, posters, staff communications and word of mouth. Patients will be enrolled following screening and consent procedures outlined below.

The research appointment will last approximately 45 - 60 minutes and include:

* Consent procedures including time for questions
* Brief interview and collection of demographic and clinical data

  * Hospital number - (for patients only)
  * Sex
  * Age
  * Ethnicity
  * Height
  * History of airway disease or surgery (including tracheostomy) or severe kyphosis of the spine
  * Major medical or surgical history will be recorded in order to provide context to clinicians reading the findings and enable them to judge applicability to their patient populations
* Measurement of weight
* Measurement of height
* Measurement of shoulder width
* Ultrasound measurement of the width of the trachea (windpipe)
* BMI will be calculated using height and weight

The following process measures will also be taken:

* Time taken to obtain measurements of the trachea
* Inter and intra-rater reliability for measurements of the trachea This information is of interest in the wider PhD programme of work. It will be presented to the Clinical Steering Committee as an indication of 1) how much time measuring the trachea would add to a tracheostomy insertion procedure and 2) accuracy of measurements.

No follow up is required after the initial research appointment. Participants may withdraw at any point up until the end of the data collection appointment. They do not have to give a reason for withdrawing and will be given assurance that their care (patients) or employment (staff) will not be affected by withdrawing. Data already collected will be kept and analysed.

The study will end when data for 114 participants have been recorded and the results described and analysed in the final study report.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 years and older) staff and patients at Royal Free London NHS Foundation Trust hospital sites (Barnet Hospital and the Royal Free Hospital).

Exclusion Criteria:

* Severe kyphosis of the spine
* Patients lacking capacity to consent
* Prisoners
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult staff and patients at the Royal Free London NHS Foundation Trust hospital sites.
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Concordance (% agreement) between size selection methods in tracheostomy | 20 months
  Concordance between 4 methods of selecting size of tracheostomy that are based on patient height, BMI, sex or shoulder width, and a method based on measurement of the trachea.

SECONDARY OUTCOMES:
Association between tracheal diameter and other patient anthropometrics/demographics | 20 months
  Strength of correlation between transverse tracheal diameter and height, shoulder width, ethnicity, age, and sex

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Newman, MSc, Principal Investigator — UCL Division of Surgery and Interventional Science (UK); Royal Free London NHS Foundation Trust (UK)
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Confidential Enquiry into Patient Outcome and Death (2014) On the right Trach? A review of the care of patients who underwent a tracheostomy. NCEPOD, London (https://www.ncepod.org.uk/2014report1/downloads/OnTheRightTrach_FullReport.pdf accessed 09/08/2021)
- [Background] Comprehensive Tracheostomy Care - The NTSP Manual [Internet]. 2013 [cited 2019 Jan 19]. p. 207. Available from: http://tracheostomy.org.uk/resources
- [Background] Bodenham, A, Bell D, Bonner S, Branch F, Dawson D, McGrath B, et al. Intensive Care Society Standards for the care of adult patients with a temporary Tracheostomy. 2014.
- [Background] Newman H, Sutt A-L, Wallace S. 0063 Choosing the size of tracheostomy tube for adults in UK intensive care units: how do we do it? J Intensive Care Soc. 2020;21(2_suppl):37-8
- [Background] De Leyn P, Bedert L, Delcroix M, Depuydt P, Lauwers G, Sokolov Y, Van Meerhaeghe A, Van Schil P; Belgian Association of Pneumology and Belgian Association of Cardiothoracic Surgery. Tracheotomy: clinical review and guidelines. Eur J Cardiothorac Surg. 2007 Sep;32(3):412-21. doi: 10.1016/j.ejcts.2007.05.018. Epub 2007 Jun 27. PMID 17588767
- [Background] Dempsey GA, Morton B, Hammell C, Williams LT, Tudur Smith C, Jones T. Long-Term Outcome Following Tracheostomy in Critical Care: A Systematic Review. Crit Care Med. 2016 Mar;44(3):617-28. doi: 10.1097/CCM.0000000000001382. PMID 26584197
- [Background] Li M, Yiu Y, Merrill T, Yildiz V, deSilva B, Matrka L. Risk Factors for Posttracheostomy Tracheal Stenosis. Otolaryngol Head Neck Surg. 2018 Oct;159(4):698-704. doi: 10.1177/0194599818794456. Epub 2018 Aug 21. PMID 30130451
- [Background] Moorhouse J, Ali T, Moorhouse T, Owens D. Poorly placed tracheostomy tubes: Effects on flow and resistance. J Intensive Care Soc. 2015 Nov;16(4):282-286. doi: 10.1177/1751143715582040. Epub 2015 Apr 22. PMID 28979432
- [Background] Norwood S, Vallina VL, Short K, Saigusa M, Fernandez LG, McLarty JW. Incidence of tracheal stenosis and other late complications after percutaneous tracheostomy. Ann Surg. 2000 Aug;232(2):233-41. doi: 10.1097/00000658-200008000-00014. PMID 10903603
- [Background] Sarper A, Ayten A, Eser I, Ozbudak O, Demircan A. Tracheal stenosis aftertracheostomy or intubation: review with special regard to cause and management. Tex Heart Inst J. 2005;32(2):154-8. PMID 16107105
- [Background] Zias N, Chroneou A, Tabba MK, Gonzalez AV, Gray AW, Lamb CR, Riker DR, Beamis JF Jr. Post tracheostomy and post intubation tracheal stenosis: report of 31 cases and review of the literature. BMC Pulm Med. 2008 Sep 21;8:18. doi: 10.1186/1471-2466-8-18. PMID 18803874
- [Background] Farzanegan R, Feizabadi M, Ghorbani F, Movassaghi M, Vaziri E, Zangi M, Lajevardi S, Shadmehr MB. An Overview of Tracheal Stenosis Research Trends and Hot Topics. Arch Iran Med. 2017 Sep;20(9):598-607. PMID 29048922
- [Background] Pang PS, Suen LK. Stressors in the ICU: a comparison of patients' and nurses' perceptions. J Clin Nurs. 2008 Oct;17(20):2681-9. doi: 10.1111/j.1365-2702.2008.02280.x. PMID 18808637
- [Background] Rotondi AJ, Chelluri L, Sirio C, Mendelsohn A, Schulz R, Belle S, Im K, Donahoe M, Pinsky MR. Patients' recollections of stressful experiences while receiving prolonged mechanical ventilation in an intensive care unit. Crit Care Med. 2002 Apr;30(4):746-52. doi: 10.1097/00003246-200204000-00004. PMID 11940739
- [Background] Khalaila R, Zbidat W, Anwar K, Bayya A, Linton DM, Sviri S. Communication difficulties and psychoemotional distress in patients receiving mechanical ventilation. Am J Crit Care. 2011 Nov;20(6):470-9. doi: 10.4037/ajcc2011989. PMID 22045144
- [Background] Bergbom-Engberg I, Haljamae H. Assessment of patients' experience of discomforts during respirator therapy. Crit Care Med. 1989 Oct;17(10):1068-72. doi: 10.1097/00003246-198910000-00021. PMID 2791570
- [Background] Wade D, Hardy R, Howell D, Mythen M. Identifying clinical and acute psychological risk factors for PTSD after critical care: a systematic review. Minerva Anestesiol. 2013 Aug;79(8):944-63. Epub 2013 Apr 5. PMID 23558761
- [Background] Happ MB. Interpretation of nonvocal behavior and the meaning of voicelessness in critical care. Soc Sci Med. 2000 May;50(9):1247-55. doi: 10.1016/s0277-9536(99)00367-6. PMID 10728845
- [Background] Griscom NT, Wohl ME. Dimensions of the growing trachea related to age and gender. AJR Am J Roentgenol. 1986 Feb;146(2):233-7. doi: 10.2214/ajr.146.2.233. PMID 3484568
- [Background] Breatnach E, Abbott GC, Fraser RG. Dimensions of the normal human trachea. AJR Am J Roentgenol. 1984 May;142(5):903-6. doi: 10.2214/ajr.142.5.903. PMID 6609569
- [Background] Gamsu G, Webb WR. Computed tomography of the trachea: normal and abnormal. AJR Am J Roentgenol. 1982 Aug;139(2):321-6. doi: 10.2214/ajr.139.2.321. PMID 6979885
- [Background] Premakumar Y, Griffin MF, Szarko M. Morphometric characterisation of human tracheas: focus on cartilaginous ring variation. BMC Res Notes. 2018 Jan 16;11(1):32. doi: 10.1186/s13104-018-3123-1. PMID 29338790
- [Background] Or DY, Karmakar MK, Lam GC, Hui JW, Li JW, Chen PP. Multiplanar 3D ultrasound imaging to assess the anatomy of the upper airway and measure the subglottic and tracheal diameters in adults. Br J Radiol. 2013 Oct;86(1030):20130253. doi: 10.1259/bjr.20130253. Epub 2013 Aug 21. PMID 23966375
- [Background] Prasad A, Yu E, Wong DT, Karkhanis R, Gullane P, Chan VW. Comparison of sonography and computed tomography as imaging tools for assessment of airway structures. J Ultrasound Med. 2011 Jul;30(7):965-72. doi: 10.7863/jum.2011.30.7.965. PMID 21705729
- [Background] Lakhal K, Delplace X, Cottier JP, Tranquart F, Sauvagnac X, Mercier C, Fusciardi J, Laffon M. The feasibility of ultrasound to assess subglottic diameter. Anesth Analg. 2007 Mar;104(3):611-4. doi: 10.1213/01.ane.0000260136.53694.fe. PMID 17312218